CLINICAL TRIAL: NCT04588272
Title: Non-invasive Carbon Dioxide Monitoring During Moderate Sedation at Different Oxygen Flow Rates in Patients Undergoing Endoscopic Retrograde Cholangio-pancreatography
Brief Title: Non Invasive End Tidal Carbon Dioxide Monitoring During Moderate Sedation
Acronym: EtCO2
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Reda Mohamed, Principal Investigator, Assiut University
Other Study IDs: Non invasive EtCO2 monitoring.
Record Dates: First submitted 2020-04-28; First posted 2020-10-19 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Carbon Dioxide
Keywords: Non invasive EtCO2 MONITORING

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2 liters: 40 patients will receive O2 supply at rate of 2 liters per minute and then cabnographic and other measures will be recorded through out the procedure.
  Interventions: Device: DualGuard
- 4 liters: 40 patients will receive receive O2 supply at rate 4 liters per minute and then cabnographic and other measures will be recorded through out the procedure.
  Interventions: Device: DualGuard
- 6 liters: : 40 patients will receive O2 supply at rate 6 liters per minute and then cabnographic and other measures will be recorded through out the procedure.
  Interventions: Device: DualGuard

INTERVENTIONS:
Device: DualGuard — DualGuard device (FlexiCare) which incorporate an endoscopy bite block with oxygen delivery and CO2 monitoring from both the mouth and nose simultaneously.

SUMMARY:
CO2 monitoring through non-invasive methods at different O2 flow rates may provide an early warning sign of hypoventilation during procedural sedation.

DETAILED DESCRIPTION:
Sedation is a drug-induced depression in the level of consciousness. The clinical objectives of administering sedation for GI endoscopy are to relieve patient anxiety and discomfort, improve the outcome of the examination, and diminish the patient's memory of the event. A number of different sedatives and analgesics can be used to achieve appropriate levels of sedation for GI endoscopic procedures. The targeted level of sedation may vary depending on patient and procedural variables, and doses of sedatives should be titrated accordingly to achieve a safe, comfortable, and technically successful endoscopic procedure. Knowledge of the pharmacologic profiles of sedation agents is necessary to maximize the likelihood that the desired level of sedation is achieved.(1) All patients receiving sedation to facilitate endoscopic procedures should have monitoring of cardiorespiratory parameters before, during, and after administration of sedation/analgesia. Electronic monitoring may detect early signs of patient distress and is an adjunct to continuous clinical assessment. Commonly used monitoring equipment for patients undergoing endoscopic procedures includes pulse oximetry, single-lead continuous electrocardiographic (ECG) monitoring, and automated blood pressure monitoring. With the increased use of propofol to facilitate endoscopy in recent years, less familiar monitoring devices have been introduced, including end-tidal carbon dioxide (EtCO2) and level of consciousness monitors. Given a recent change in the American Society of Anesthesiologists (ASA) guidelines, recommending CO2 monitoring for patients undergoing both moderate and deep sedation, familiarity with capnography may become necessary.(2) Patients are at risk of respiratory depression and acute hypercapnia during sedation and recovery from anaesthesia . Desaturation on pulse oximetry for monitoring of hypoventilation is a late sign. Moreover, hypoventilation is masked by administration of supplemental O2. ( 3) For a sedated patient in spontaneous ventilation, hypoventilation (by airway obstruction or central respiratory depression) will likely precede hypoxemia. Hence, if the patient is monitored using a capnograph machine, when hypoventilation occurs, PEtCO2 increases and the shape of the capnography curve is modified.This may trigger an adequate response from the person monitoring the anesthesia (chin thrust, sedative dose modification, oxygen supplementation) so as to prevent hypoxemia. (5) Measuring CO2 noninvasively includes capnography and capnometry. capnography provides numerical and graphical (waveforms) forms, while capnometry provides only numerical form. (6) Arterial blood gas (ABG) can tell us about the patient's acid-base balance, which is measured by the hydrogen ion (H) concentration in the blood (pH), oxygen saturation (SaO2), partial pressure of oxygen (PaO2), partial pressure of carbon dioxide (PaCO2), concentration of bicarbonate (HCO3), base excess and base deficit.(7) ABG results can indicate how effectively the patient's body is compensating for the acid-base disturbance and whether the patient's total blood volume is adequate for transporting all the nutrients that the body's tissues require. (8)

Hyopthesis of this trial: is CO2 monitoring through non-invasive methods may provide an early warning sign of hypoventilation during procedural sedation.

Primary outcome: Measuring end-tidal carbon dioxide (EtCO2) that is taken during different flows of oxygen(O2) supplementation.

Secondary outcome: Will include O2 saturation, haemodynamics (systolic blood pressure, diastolic blood pressure and mean blood pressure), time to recovery, patient satisfaction, Ramsay sedation scale (which is used to measure level of sedation through dividing patients level of sedation into 6 categories ranging from severe agitation to deep coma). (9) Ramsay Sedation Scale

1. Patient is anxious and agitated or restless, or both.
2. Patient is co-operative, oriented, and tranquil.
3. Patient responds to commands only.
4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
6. Patient exhibits no response.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult Patients aged 20-60 years.
* Sex: either male or female.
* ASA physical status I or II.
* Elective ERCP

Exclusion Criteria:

* Abnormal renal function test.
* History of asthma or COPD
* patients with a history of hypertension and diabetes.
* Cardiac patients.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: : Two days before surgery, patients will visit the outpatient clinic for history taken, clinical assessment and explanation about the study protocol. Laboratory investigations will be performed and patients will be informed that they can stop participation in the study at any time without any loss of service.
  Patients will receive conscious sedation via propofol 1.5 mg/kg and lidocaine 1 mg/kg and CO2 monitored through non-invasive method.
  At the end of the procedure, all patients will recover until full consciousness regains and they are able to follow verbal commands. After the desired spontaneous ventilation, the patients will be transferred to the recovery room.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
End-tidal carbon dioxide | During the procedure.
  : end-tidal carbon dioxide (EtCO2) that is taken during different flows of oxygen(O2) supplementation will be measured.

SECONDARY OUTCOMES:
Oxygen saturation. | During the procedure.
  : Measuring O2 saturation at different O2 flow rates.
Haemodynamics as blood pressure. | During the procedure.
  Measuring systolic blood pressure, diastolic blood pressure and mean blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fathy, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt